CLINICAL TRIAL: NCT06660199
Title: Effectiveness of Text-based Support for Parents of Suicidal Adolescents Following Emergency Department Visits
Brief Title: Text-based Support for Parents of Adolescents Following an Emergency Department Visits
Acronym: TESP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Ewa Czyz, Associate Professor of Psychiatry, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HUM00254540; 1R01MH137012-01 (NIH)
Record Dates: First submitted 2024-10-23; First posted 2024-10-28 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Suicide
Keywords: Text; Suicidal Ideation; Suicide Attempt
MeSH Terms: conditions — Suicide; Suicidal Ideation; Suicide, Attempted

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard ED care (No Intervention)
- Standard ED care with a text-based intervention (Experimental): This arm incorporates adolescent-centered (A-C) and parent-centered (P-C) texting components
  Parents in the intervention arm will receive up to 3 text messages per day over six weeks after ED discharge: daily A-C text and up to two P-C messages. The P-C component includes an embedded micro-randomized trial (MRT), and parents will be randomized twice each day over the six-week intervention to either receive or not receive a P-C message.
  Interventions: Behavioral: Text-based intervention

INTERVENTIONS:
Behavioral: Text-based intervention — Parents randomized to the texting intervention will receive up to 3 messages each day for 6 weeks: The intervention is comprised of adolescent-centered (A-C) texts focusing on parental adherence to recommended suicide prevention strategies to promote adolescents' safety and parent-centered (P-C) texts focused on improving parents' own well-being.
  Arms: Standard ED care with a text-based intervention

SUMMARY:
The goal of this study is to determine the effectiveness of an adaptive text-based intervention for parents of adolescents seeking emergency department services for suicide risk concerns.

DETAILED DESCRIPTION:
Participants will be 420 adolescents (ages 13-17) seen in ED with recent suicidal ideation and/or attempt and their parents recruited from two health system EDs in the Midwest.

ELIGIBILITY:
Inclusion Criteria:

* Adolescent (13-17 years old) who present to Emergency Department (ED) due to (1) last-week suicidal ideation and/or (2) last-month suicide attempt, and their caregiver.

Exclusion Criteria:

Adolescents who are:

* medically unstable
* presenting with severe cognitive impairment, altered mental status, severe aggression/agitation
* presenting without a legal guardian
* whose parent does not own a cell phone

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 420 (Estimated)
Dates: Start 2025-12-01 (Actual); Primary Completion 2028-07 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Aim 1 (primary aim): likelihood of suicidal behavior (actual, interrupted, or aborted attempts) | 12-week follow-up
  Suicidal behavior encompasses actual, interrupted, and aborted suicide attempts. Measured with the behavioral subscale of the Columbia-Suicide Severity Rating Scale (C-SSRS),and supplemented with available medical chart data.
Aim 2 (secondary aim) severity of parental stress | Up to 6 weeks
  Measured with twice daily surveys over the 6-week intervention

SECONDARY OUTCOMES:
Aim 1 (primary aim): -time- to- suicidal behavior (actual, interrupted, or aborted suicide attempts | 24-week follow-up
  Measured with the behavioral subscale of C-SSRS and supplemented with available chart data.
Aim 1 (primary aim): time- to- return ED visit | 24-week follow-up.
Aim 2 (secondary aim): parental negative affect | Up to 6 weeks
  Measured with twice daily surveys over the 6-week intervention.
Aim 2 (secondary aim) parental positive affect | Up to 6 weeks
  Measured with twice daily surveys over the 6-week intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Ewa Czyz, Ph.D., Principal Investigator — University of Michigan
Locations (2):
- United States (2):
  - University of Michigan, Ann Arbor, Michigan
  - Hurley Medical Center, Flint, Michigan

IPD SHARING:
Plan to Share IPD: No